CLINICAL TRIAL: NCT04570891
Title: Ultrasound-guided Fascia Iliaca Compartment Block for Proximal Femoral Osteotomy in Pediatric Patients: a Randomized Controlled Trial
Brief Title: Ultrasound-guided FICB for Proximal Femoral Osteotomy in Pediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2008-003-1145
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FICB (Experimental): Ultrasound-guided fascia iliaca compartment block (0.25% ropivacaine 1mL/kg, Max 30mL) will be provided at the end of surgery.
  Interventions: Procedure: Ultrasound-guided fascia iliaca compartment block
- Control (Placebo Comparator): No regional block is provided at the end of surgery.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Ultrasound-guided fascia iliaca compartment block — Ultrasound-guided fascia iliaca compartment block (0.25% ropivacaine 1mL/kg, Max 30mL) will be provided at the end of surgery.
  Arms: FICB
Procedure: Control — No regional block is provided at the end of surgery.
  Arms: Control

SUMMARY:
This prospective randomized controlled trial aims to examine the effect of fascia iliaca compartment block on the postoperative pain and opioid consumption in pediatric patients (3y≤ age <18y) who will undergo orthopedics surgery (proximal femoral osteotomy).

Patients will be allocated to either the FICB(Fascia iliaca compartment block + IV PCA) group or the control group (no block + IV PCA). Fascia iliaca compartment block will be performed using 0.25% ropivacaine (1mL/kg, MAX 30mL) under ultrasound-guidance at the end of surgery.

The total opioid consumption at 12, and 24 hours after the surgery, and the pain score at 10 min after PACU admin, 1,6,24 hours after the surgery, the total dose of additional rescue analgesia (intravenous ketorolac or nalbuphine) at 12 and 24 hours after the surgery will be recorded.

DETAILED DESCRIPTION:
This prospective randomized controlled trial aims to examine the effect of fascia iliaca compartment block on postoperative pain and opioid consumption in pediatric patients (3y≤ age <18y) who will undergo orthopedics surgery (proximal femoral osteotomy).

Patients will be allocated to either the FICB(Fascia iliaca compartment block + IV PCA) group or the control group (no block + IV PCA). Fascia iliaca compartment block will be performed using 0.25% ropivacaine (1mL/kg, MAX 30mL) under ultrasound-guidance at the end of surgery.

The total opioid consumption at 12, and 24 hours after the surgery, and the pain score at 10 min after PACU admin, 1,6,24 hours after the surgery, the total dose of additional rescue analgesia (intravenous ketorolac or nalbuphine) at 12 and 24 hours after the surgery will be recorded.

ELIGIBILITY:
Inclusion Criteria:

- 36 children aged between 3 and 18 years who undergo proximal femoral osteotomy

Exclusion Criteria:

* Complex surgery (other than proximal femoral osteotomy)
* Allergy to opioid
* Allergy to local anesthetics
* Disease in heart, lung, kidney, and liver
* Coagulation disorder
* Disease in the central and peripheral nervous system
* Unstable vital sign
* Significant renal impairment (Creatinine> 3.0 mg/dl)
* Significant hepatic impairment (aspartate transaminase> 120 unit/L, alanine aminotransferase> 120 unit/L)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
total opioid consumption at 12 hours after the end of surgery | at 12 hours after the end of surgery
  total opioid consumption at 12 hours after the end of surgery (IV Nalbuphine 1mg = IV Morphine 1mg = IV Fentanyl 10mcg (0.01mg) per kilogram of body weight.

SECONDARY OUTCOMES:
total opioid consumption at 24 hours after the end of surgery | at 24 hours after the end of surgery
  total opioid consumption at 24 hours after the end of surgery (IV Nalbuphine 1mg = IV Morphine 1mg = IV Fentanyl 10mcg (0.01mg) per kilogram of body weight.
Wong-Baker Faces Pain Rating Scale | at 10 minutes after the PACU admin, 1hour, 6hours, and 24hours after the end of surgery.
  by Wong-Baker Faces Pain Rating Scale: There are 6 faces in the Wong-Baker Pain Scale. The first face represents a pain score of 0, and indicates "no hurt". The second face represents a pain score of 2, and indicates "hurts a little bit." The third face represents a pain score of 4, and indicates "hurts a little more". The fourth face represents a pain score of 6, and indicates "hurts even more". The fifth face represents a pain score of 8, and indicates "hurts a whole lot"; the sixth face represents a pain score of 10, and indicates "hurts worst".
Numeric rating scale | 10 minutes after the PACU admin, 1hour, 6hours, and 24hours after the end of surgery.
  by Numeric rating scale: A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable.
Total additional dose of nalbuphine | at 12hours, and 24hours after the end of surgery.
  Total additional dose of nalbuphine (mg) per kilogram of body weight.
Total additional dose of ketorolac | at 12hours, and 24hours after the end of surgery.
  Total additional dose of ketorolac (mg) per kilogram of body weight.
The incidence of side effects of analgesic medications | within 24 hours after the end of surgery
  Nausea, Vomit, Constipation, Pruritus, Dizziness, Dry mouth, Sedation
The incidence of side effects of ropivacaine | within 1 hour after the end of surgery
  Arrhythmia, Hypotension, ST change, Dizziness, Convulsion
Hospital stay | within 14 days after the end of surgery
  Hospital stay (days)
Neurological Pupil indexTM (NPi) | at 1 hour after the end of surgery
  measured by pupillometer
pupil constriction velocity (CV) | at 1 hour after the end of surgery
  measured by pupillometer
Extensor hallucis longus function (motor power of extension of the big toe: I-V) at the second postoperative day (POD-2) | At the second postoperative day (POD-2)
  Extensor hallucis longus function (motor power of extension of the big toe: I-V) at the second postoperative day (POD-2)
Intact toe sensory at the second postoperative day (POD-2) | At the second postoperative day (POD-2)
  Intact toe sensory at the second postoperative day (POD-2)
Normal capillary refill time (< 3 seconds) at the second postoperative day (POD-2) | At the second postoperative day (POD-2)
  Normal capillary refill time (< 3 seconds) at the second postoperative day (POD-2)

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided